CLINICAL TRIAL: NCT04941820
Title: The Impact of Clinical Pharmacist in the Identification and Management of Treatment Related Problems in the Surgery Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hiba Al Fahmawi, Study Director, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80/2019/1943
Record Dates: First submitted 2021-06-08; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Surgical Patients
Keywords: clinical pharmacist; general surgical ward; RCT; SICU

STUDY DESIGN:
Intervention Model Description: All patients were followed up prospectively for their length of hospital stay, and recommendations concerning each identified TRP were provided to the surgeons responsible for patients in the intervention group. Likewise, patient counseling and encouraging adherence to therapy were provided solely to patients in the intervention group. Patients in the control group received usual care by the surgical team without a coordinated contribution from the clinical pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical pharmacist intervention + usual care arm (Experimental): Patients in the clinical pharmacist intervention + usual care arm received the clinical pharmacist intervention as well as usual care provided by the surgical team
  Interventions: Other: clinical pharmacist intervention
- Usual care arm (Control arm) (No Intervention): Patients in the control arm received usual care by the surgical team without a coordinated contribution from the clinical pharmacist

INTERVENTIONS:
Other: clinical pharmacist intervention — clinical pharmacist intervention
  Arms: Clinical pharmacist intervention + usual care arm

SUMMARY:
Patients in the surgery ward are at risk of morbidity and mortality from various types of treatment-related problems (TRPs). The primary aim of this study is to assess the impact of the clinical pharmacist in the identification and management of TRPs in the surgery ward.

DETAILED DESCRIPTION:
Patients were randomly assigned to intervention (n=50) and usual care (n=50) arms. The clinical pharmacist assessed the types, frequencies, and clinical significance of TRPs for all recruited patients at baseline. Patients and treating surgeons in the intervention arm received recommendations concerning the identified TRPs, while the usual care arm did not. The number of TRPs was reevaluated at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Admission for elective, urgent, or emergency surgery
* age 18 years or older
* Expected length of stay of 3 days or more in the general surgical ward or the SICU

Exclusion Criteria:

* Pregnancy, breastfeeding, drug or alcohol abuse, active malignancy, or admission for plastic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of clinical pharmacist's recommended interventions | 19-week
  (Number of recommendations accepted by surgeons) / (total number of recommendations submitted to surgeons by the clinical pharmacist) *100
Implementation rate of clinical pharmacist's recommended interventions | 19-week
  (Number of recommendations implemented by surgeons and patients) / (total number of recommendations submitted to surgeons and patients by the clinical pharmacist) *100
The impact of the clinical pharmacist on the identification and management of TRPs in the surgery ward | 19-week
  Measured by comparing the means of differences in the number of TRPs identified at baseline and at the time of short-term follow-up in the intervention and usual care groups

SECONDARY OUTCOMES:
Surgeons' attitudes and satisfaction towards the provided clinical pharmacy services | 19-week
  Measured by a self-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hiba I. Al Fahmawi, PharmD, MSc, Study Director — School of Pharmacy, The University of Jordan, Amman, Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Background] AbuRuz SM, Bulatova NR, Yousef AM. Validation of a comprehensive classification tool for treatment-related problems. Pharm World Sci. 2006 Aug;28(4):222-32. doi: 10.1007/s11096-006-9048-0. Epub 2006 Oct 26. PMID 17066238
- [Background] Basheti IA, Ayasrah SM, Ahmad M. Identifying treatment related problems and associated factors among hospitalized post-stroke patients through medication management review: A multi-center study. Saudi Pharm J. 2019 Feb;27(2):208-219. doi: 10.1016/j.jsps.2018.10.005. Epub 2018 Oct 19. PMID 30766431
- [Background] Bilal AI, Tilahun Z, Beedemariam G, Ayalneh B, Hailemeskel B, Engidawork E. Attitude and satisfaction of health care providers towards clinical pharmacy services in Ethiopia: A post-deployment survey. J Pharm Policy Pract. 2016 Mar 8;9:7. doi: 10.1186/s40545-016-0058-6. eCollection 2016. PMID 26962456
- [Background] Hepler CD. Clinical pharmacy, pharmaceutical care, and the quality of drug therapy. Pharmacotherapy. 2004 Nov;24(11):1491-8. doi: 10.1592/phco.24.16.1491.50950. PMID 15537552